CLINICAL TRIAL: NCT06669208
Title: A Double Blind, Randomized, Placebo-Controlled, Phase 1 Dose Escalation Trial to Evaluate the Safety and Immunogenicity of an Inactivated Chikungunya Virus Vaccine, HydroVax-005 CHIKV, in Healthy Adults
Brief Title: Trial of an Inactivated Chikungunya Virus Vaccine
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Najit Technologies, Inc. (Industry)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Prevention
Other Study IDs: 24-0001; U44AI152995 (NIH)
Record Dates: First submitted 2024-10-30; First posted 2024-11-01 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Chikungunya Fever; Chikungunya Virus; Chikungunya
Keywords: Chikungunya virus; HydroVax; dose-ranging; double blind; placebo-controlled; vaccine
MeSH Terms: conditions — Chikungunya Fever

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Low Dose (Experimental): 20 subjects will receive 2.5 mcg intramuscularly (IM) of HydroVax-005 CHIKV on Days 1 and 29
  Interventions: Biological: HydroVax-005 CHIKV
- High Dose (Experimental): 20 subjects will receive 8 mcg intramuscularly (IM) of HydroVax-005 CHIKV on Days 1 and 29
  Interventions: Biological: HydroVax-005 CHIKV
- Placebo (Placebo Comparator): 8 subjects will receive normal saline placebo intramuscularly (IM) on Days 1 and 29
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: HydroVax-005 CHIKV — HydroVax-005 CHIKV vaccine
  Arms: High Dose; Low Dose
Other: Placebo — NaCl 0.9%, Normal Saline
  Arms: Placebo

SUMMARY:
This trial will be a randomized, placebo controlled, double-blind (within dosing group), dose escalation Phase 1 trial, evaluating dosages of 2.5 mcg and 8 mcg of HydroVax-005 CHIKV vaccine given intramuscularly on Day 1 and Day 29 in up to 48 healthy adults healthy adults ≥ 18 and < 50 years of age. The primary objective is to assess the safety and reactogenicity of the HydroVax-005 CHIKV vaccine administered intramuscularly in a two-dose series on Days 1 and 29 at a dose of 2.5 mcg or a dose of 8 mcg.

DETAILED DESCRIPTION:
This trial will be a randomized, placebo controlled, double-blind (within dosing group), dose escalation Phase 1 trial evaluating dosages of 2.5 mcg and 8 mcg of HydroVax-005 CHIKV vaccine given intramuscularly on Day 1 (the day of first vaccination is defined as Day 1) and Day 29 in healthy adults ≥ 18 and < 50 years of age. The study will consist of two dosing groups of HydroVax-005 CHIKV vaccine to be enrolled sequentially. Each dose group will consist of 20 individuals who receive HydroVax-002 YFV, as well as 8 total subjects who receive placebo. Each dose-group will include a sentinel subgroup consisting of 5 vaccine and 1 placebo recipient. In each of the two (2.5 mcg and 8 mcg) dose phases, enrollment is halted after the dose 1 vaccination of the sentinel subgroup. Following assessment of safety and reactogenicity data of Group 1 by the Internal Safety Review Committee (ISRC), the vaccine dose will be increased to 8 mcg for Group 2.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent prior to initiation of any study procedures.
2. Are able to understand and comply with planned study procedures and be available for all study visits.
3. Must agree to the collection of venous blood per protocol.
4. Are males or non-pregnant females, ≥18 and <50 years of age, inclusive at time of enrollment.
5. Are in good health. As determined by medical history and physical examination to evaluate acute or currently ongoing chronic medical or psychiatric diagnoses or conditions, defined as those that have been present for at least 90 days, which would affect the assessment of the safety of subjects or the immunogenicity of study vaccinations. Chronic medical diagnoses or conditions should be stable for the last 60 days (no hospitalizations, emergency room or urgent care for condition, or invasive medical procedure and no adverse symptoms that need medical intervention such as medication change/supplemental oxygen). This includes no change in chronic prescription medication, dose or in the 60 days prior to enrollment. Any prescription change that is due to change of health care provider, insurance company, etc., or that is done for financial reasons, as long as in the same class of medication, will not be considered a deviation of this inclusion criterion. Subjects may be on chronic or as needed (prn) medications if, in the opinion of the site PI or appropriate sub-investigator, they pose no additional risk to subject safety or assessment of reactogenicity and immunogenicity and do not indicate a worsening or treatment of continued symptoms of medical diagnosis or condition. Note: Low dose topical, corticosteroids as outlined in the Subject Exclusion Criteria as well as herbals, vitamins and supplements are permitted.
6. Oral temperature is less than 100.0℉.
7. Pulse is 40 to 100 beats per minute, inclusive.
8. Systolic blood pressure is 90 to 140 mmHg, inclusive.
9. Diastolic blood pressure is 60 to 90 mmHg, inclusive.
10. Screening laboratories (White Blood Cell Count (WBC), Hemoglobin (Hgb), Platelet Count (PLTs), Sodium, Potassium, Bicarbonate, Calcium, Creatinine (Cr), Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST), Total Bilirubin (TBIL) and urine protein and glucose) are within acceptable parameters. Hematology, blood chemistry and liver enzymes must be Grade 1 or less at screening; urine glucose negative and urine protein no greater than trace at screening for subjects to qualify for randomization and vaccination.
11. Negative test result at screening blood draw for hepatitis B virus (HBV) surface antigen (HBsAg), hepatitis C virus (HCV) antibody or human immunodeficiency virus (HIV) types 1 or 2 antibodies.
12. Women of childbearing potential must use an acceptable contraception method from at least 30 days before the first study vaccination until 30 days after the second study vaccination. Not sterilized via, bilateral oophorectomy, salpingectomy, hysterectomy, or successful Essure® placement (permanent, non-surgical, non-hormonal sterilization) with documented radiological confirmation test at least 90 days after the procedure, and still menstruating or <1 year has passed since the last menses if menopausal. Includes non-male sexual relationships, full abstinence from sexual intercourse with a male partner, monogamous relationship with vasectomized partner who has been vasectomized for 180 days or more and shown to be azoospermic prior to the subject receiving the study vaccination, effective intrauterine devices, NuvaRing®, tubal ligation, and licensed hormonal methods such as implants, injectables or oral contraceptives (i.e. "the pill").
13. Women of childbearing potential must have a negative serum pregnancy test at screening and a negative urine pregnancy test within 24 hours prior to each study vaccination.
14. Sexually active males must agree to use a medically acceptable form of contraception in order to be in this study and must agree to continue such use until day 90 after the last vaccination. Medically acceptable contraceptives include: (1) surgical sterilization (such as a vasectomy), or (2) a condom used with a spermicide. Contraceptive measures such as Plan B™, sold for emergency use after unprotected sex, are not acceptable methods for routine use.

Exclusion Criteria:

1. Have an acute illness or acute febrile illness (oral temperature ≥ 38℃ [100.4℉]), as determined by the site PI or appropriate sub-investigator, within 72 hours prior to study vaccination. An acute illness which is nearly resolved with only minor residual symptoms remaining is allowable if, in the opinion of the site PI or appropriate sub-investigator, the residual symptoms will not interfere with the ability to assess safety parameters as required by the protocol.
2. Have any medical disease or condition that, in the opinion of the site PI or appropriate sub-investigator, is a contraindication to study participation. Including acute, subacute, intermittent or chronic medical disease or condition that would place the subject at an unacceptable risk of injury, render the subject unable to meet the requirements of the protocol, or may interfere with the evaluation of responses or the subject's successful completion of this trial.
3. Have immunosuppression as a result of an underlying illness or treatment, a recent history or current use of immunosuppressive or immunomodulating disease therapy.
4. Use of anticancer chemotherapy or radiation therapy (cytotoxic) within 3 years prior to study vaccination.
5. Have known active or recently active (12 months) neoplastic disease or a history of any hematologic malignancy. Non-melanoma, treated, skin cancers are permitted.
6. Known allergy to components of the study product. Including the following: aluminum hydroxide, sorbitol, potassium chloride, sodium chloride and polysorbate80 (Tween80)
7. Unstable seizure disorder (defined as requiring medication for seizure control or with seizure activity within the past 3 years).
8. Have a history of alcohol or drug abuse within 5 years prior to study vaccination.
9. Have any diagnosis, current or past, of schizophrenia, bipolar disease or other psychiatric diagnosis that may interfere with subject compliance or safety evaluations. As determined by the site PI or appropriate sub-investigator.
10. Have been hospitalized for psychiatric illness, history of suicide attempt, or confinement for danger to self or others within 5 years prior to study vaccination.
11. Have a history of asthma, other than mild, well-controlled asthma. Cold or exercise induced asthma controlled with inhaled medications other than inhaled corticosteroids is permissible. Participants should be excluded if they require daily bronchodilator use, or have had an asthma exacerbation requiring oral/parenteral steroid use or have used theophylline or inhaled corticosteroids in the past year.
12. Have a history of diabetes mellitus.
13. Have taken oral or parenteral (including intra-articular) or chronic topical corticosteroids of any dose within 30 days prior to study vaccination. Corticosteroid nasal sprays for allergic rhinitis are permissible. Persons using a topical corticosteroid for a limited duration for mild uncomplicated dermatitis such as poison ivy or contact dermatitis may be enrolled the day after their therapy is completed.
14. Have taken high-dose inhaled corticosteroids within 30 days prior to study vaccination. High-dose defined as per age as using inhaled high-dose per reference chart in the National Heart, Lung and Blood Institute Guidelines for the Diagnosis and Management of Asthma (EPR-3) or other lists published in UPTODATE.
15. Received or plan to receive a licensed, authorized or unlicensed, live vaccine within 30 days before or after each study vaccination.
16. Received or plan to receive a licensed, authorized or unlicensed, inactivated vaccine or allergy desensitization shot within 14 days before or after each study vaccination.
17. Received an experimental agent within 30 days prior to the study vaccination or expect to receive another experimental agent during the trial-reporting period. Including, drug, biologic, device, blood product, or medication.
18. Are participating or plan to participate in another clinical trial with an interventional agent that will be received during the trial-reporting period. Including licensed or unlicensed, drug, biologic, device, blood product, or medication.
19. Female subjects who are breastfeeding or plan to breastfeed from the time of the first study vaccination through 30 days after the last study vaccination.
20. Receipt of blood products or immunoglobulin within six months prior to enrollment.
21. Donation of a unit of blood within 60 days prior to enrollment or intends to donate blood during the study period.
22. Body mass index (BMI) ≥ 35.
23. History of a visit to, or prior residence in, South America, sub-Saharan Africa or Southeast Asia lasting one month or more.
24. Planned travel to areas known to be endemic with chikungunya virus during the study period.
25. History of vaccination against chikungunya virus.
26. History of vaccination with other alphavirus candidate vaccines.
27. History of chikungunya virus infection.
28. Plan to have a major change in exercise routine or perform strenuous exercise from 72 hours before any dose of study vaccine/placebo and for 72 hours before any safety laboratories. Safety laboratories are obtained on Days 4 and 15 following each dose of study product.
29. Contraindication to intramuscular vaccination of either upper arm (for example, due to lymphadenectomy or obscuring tattoos).
30. History of chronic arthralgia or arthritis

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-11-04 (Actual); Primary Completion 2026-02-20 (Estimated); Study Completion 2026-02-20 (Estimated)

PRIMARY OUTCOMES:
Occurrence of all serious adverse events (SAEs) at any time during the study | Day 1 post first vaccination to Day 180 post second vaccination
  Occurrence of all serious adverse events (SAEs) at any time during the study
Incidence of Adverse Events of Special Interest (AESI) at any time during the study | Day 1 post first vaccination to Day 180 post second vaccination
  Incidence of Adverse Events of Special Interest (AESI) at any time during the study
Occurrence of all Grade 3 unsolicited adverse events (AEs) from first vaccination through day 29 after the second vaccination | Through day 29 after the second vaccination
  Occurrence of all Grade 3 unsolicited adverse events (AEs) from first vaccination through day 29 after the second vaccination
Occurrence of all Grade 3 laboratory toxicities from first vaccination through day 15 after the second vaccination | Through day 15 after the second vaccination
  Occurrence of all Grade 3 laboratory toxicities from first vaccination through day 15 after the second vaccination
Occurrence of solicited local AE and reactogenicity signs and symptoms in the 7 days after each vaccination | Through 7 days after each vaccination
  Occurrence of solicited local AE and reactogenicity signs and symptoms in the 7 days after each vaccination
Occurrence of solicited systemic AE and reactogenicity signs and symptoms in the 7 days after each vaccination | Through 7 days after each vaccination
  Occurrence of solicited systemic AE and reactogenicity signs and symptoms in the 7 days after each vaccination
Occurrence of any AE through day 29 after the second vaccination | Through day 29 after the second vaccination
  Occurrence of any AE through day 29 after the second vaccination

SECONDARY OUTCOMES:
Percentage of subjects achieving seroconversion | At day 29 after first vaccination and at day 29 after second vaccination
  Percentage of subjects achieving seroconversion (≥1:10 in plaque reduction neutralizing titer [PRNT50] titer, at day 29 after first vaccination and at day 29 after second vaccination
Geometric mean neutralizing titers | At days 15 and 29 after first vaccination and at days 15, 29, 57, and 180 following second vaccination
  Geometric mean neutralizing titers at days 15 and 29 after first vaccination and at days 15, 29, 57, and 180 following second vaccination
Reverse cumulative distribution curve of neutralizing titers | At days 15 and 29 after first vaccination and at days 15, 29, 57, and 180 following second vaccination
  Reverse cumulative distribution curve of neutralizing titers on Days 15 and 29 after first vaccination and at days 15, 29, 57, and 180 after the second vaccination for each dose group and for all dose groups combined

CONTACTS AND LOCATIONS:
Locations (1):
- Duke University Health System, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided